CLINICAL TRIAL: NCT02328846
Title: Transcutaneous-Arterial Carbon Dioxide Gradient Predicts Microcirculatory Dysfunction And The Development of Organ Failure After Cardiac Surgery
Brief Title: Transcutaneous-Arterial Carbon Dioxide and Microcirculatory Dysfunction
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient equipment
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Bhiken I. Naik, MD, Assistant Professor, University of Virginia
Other Study IDs: 17872
Record Dates: First submitted 2014-12-18; First posted 2014-12-31 (Estimated); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Bypass Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Evaluation of the microcirculation is currently limited. Continual assessment of the tissue carbon dioxide-arterial carbon dioxide (PtC02-aCO2) offers a new, novel and noninvasive method of determining the state of the microcirculation. The investigators will apply two non-invasive devices, the Braedius sidesteam darkfield microscopy (SDF) microscopy device to the sublingual circulation and the transcutaneous PtC02 probe to the forehead in subjects undergoing cardiac surgery with cardiopulmonary bypass. The PtC02-aCO2 gradient will be determined and correlated with the videomicroscopic images of the sublingual microcirculation. Thereafter the incidence of postoperative organ failure and acute kidney injury will be determined and correlated with PtC02-arterial CO2 gradient and videomicroscopic images.

Data will be analyzed by standard descriptive statistical methods.

DETAILED DESCRIPTION:
There is increasing evidence that despite resuscitation and normalization of macrohemodynamic parameters (blood pressure and cardiac output) significant dysfunction of the microcirculation may persist.1, 2 There is also a positive correlation between the severity of microcirculatory dysfunction and outcome in patients with septic shock. In contrast, early improvements in microcirculatory perfusion in response to macrohemodynamic goal directed therapy is associated with an improvement in organ function.3 Monitoring the microcirculation is challenging. The monitoring window (e.g. the sublingual bed) must be reflective of other remote vascular beds. This is more likely to be the case in the setting of systemic diseases such as sepsis and hypovolemic shock. Current research modalities for studying the microcirculation include laser Doppler and videomicroscopy.4 The limitation of these devices is that assessment of the microcirculation has to be performed off-line and targets for microvascular resuscitation have not been established. Therefore, microvascular monitoring is currently restricted to the research arena. Evaluation of the tissue transcutaneous carbon dioxide (PtC02) is a novel, non-invasive, real-time method of assessing the microcirculation.5, 6 The three major determinants of PtC02 are arterial carbon dioxide (PaCO2), oxygen consumption (VCO2) and the tissue blood flow. Under normal conditions, an increased tissue metabolism (thus VCO2) is coupled with an increased tissue perfusion, largely reducing any PtC02 increase ("washout" phenomenon). Therefore, if PaCO2 is constant, an increase in PtC02 reflects an inadequate relationship between metabolism and tissue perfusion. PtC02 thus represents a good estimate of tissue perfusion. To overcome the influence of PaCO2 on PtC02, it is convenient to use the carbon dioxide gap (tissue-arterial carbon dioxide gradient, normal<7 mmHg). Very high gap values may in addition suggest the presence of tissue hypoxia while moderately elevated gaps may represent either flow stagnation or tissue hypoxia. Cardiac surgery is characterized by significant alteration of the microvascular circulation. These changes are observed in both on-pump and off-pump cases and with pulsatile and non-pulsatile flow. Monitoring the PtC02-arterial CO2 gradient offers a rapid real-time measure of the microvascular abnormalities encountered during the post-cardiopulmonary bypass (CPB) period and their effect on post-CPB organ dysfunction.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Elective cardiac surgery
3. Must be able to read and speak English

Exclusion Criteria:

1. Subjects unable/unwilling to give informed consent
2. Emergency surgery
3. Age < 18 years
4. Pregnant females-self reported
5. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing cardiac surgery with cardiopulmonary bypass
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-01 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Postoperative SOFA score | Participants will be followed for the duration of ICU stay, an expected average of 1 weeks

SECONDARY OUTCOMES:
Postoperative Kidney Disease Improving Global Outcome (KDIGO) class | Participants will be followed for the duration of ICU stay, an expected average of 1 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Bhiken I Naik, M.B.B.Ch, Principal Investigator — University of Virginia

REFERENCES:
- [Result] Asfar P, Meziani F, Hamel JF, Grelon F, Megarbane B, Anguel N, Mira JP, Dequin PF, Gergaud S, Weiss N, Legay F, Le Tulzo Y, Conrad M, Robert R, Gonzalez F, Guitton C, Tamion F, Tonnelier JM, Guezennec P, Van Der Linden T, Vieillard-Baron A, Mariotte E, Pradel G, Lesieur O, Ricard JD, Herve F, du Cheyron D, Guerin C, Mercat A, Teboul JL, Radermacher P; SEPSISPAM Investigators. High versus low blood-pressure target in patients with septic shock. N Engl J Med. 2014 Apr 24;370(17):1583-93. doi: 10.1056/NEJMoa1312173. Epub 2014 Mar 18. PMID 24635770
- [Result] De Backer D, Creteur J, Preiser JC, Dubois MJ, Vincent JL. Microvascular blood flow is altered in patients with sepsis. Am J Respir Crit Care Med. 2002 Jul 1;166(1):98-104. doi: 10.1164/rccm.200109-016oc. PMID 12091178
- [Result] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Result] Vallee F, Mateo J, Dubreuil G, Poussant T, Tachon G, Ouanounou I, Payen D. Cutaneous ear lobe Pco(2) at 37 degrees C to evaluate microperfusion in patients with septic shock. Chest. 2010 Nov;138(5):1062-70. doi: 10.1378/chest.09-2690. Epub 2010 May 14. PMID 20472858
- [Result] Vallee F, Vallet B, Mathe O, Parraguette J, Mari A, Silva S, Samii K, Fourcade O, Genestal M. Central venous-to-arterial carbon dioxide difference: an additional target for goal-directed therapy in septic shock? Intensive Care Med. 2008 Dec;34(12):2218-25. doi: 10.1007/s00134-008-1199-0. Epub 2008 Jul 8. PMID 18607565